CLINICAL TRIAL: NCT07251270
Title: Effect of Stress Ball on Pain, Anxiety Levels, and Hemodynamic Variables During Chest Tube Removal After Open Heart Surgery
Brief Title: Effect of Stress Ball During Chest Tube Removal After Open Heart Surgery
Acronym: Stress ball
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mersin University (Other)
Collaborators: Mersin University, School of Medicine (Unknown)
Responsible Party: Principal Investigator, Tugba CAM YANIK, Assistant Professor of Surgical Diseases Nursing, Mersin University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Mersin_Unı; Tuğba ÇAM YANIK (Other: Mersin University)
Record Dates: First submitted 2025-09-16; First posted 2025-11-26 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Pain; Hemodynamic Changes; Anxiety
MeSH Terms: conditions — Pain; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: single blind
Who Masked: Outcomes Assessor
Masking Description: Since only patients in the study group will be administered, the study will not be blinded. Upon completion of the study, data from the study and control groups (coded as A or B) will be transferred to a computer by a researcher independent of the study, and the data will be analyzed and reported using a blinded technique by a statistician. Therefore, the study will be conducted as a single-blind clinical trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (No Intervention): Chest tubes are routinely removed on the second or third postoperative day in patients in the Cardiovascular Surgery Intensive Care Unit, and patients with stable hemodynamic variables are discharged to the clinic. Morphine (0.01 mg) and paracetamol (if necessary) are used for routine analgesic treatment during the intensive care unit. Data will be collected between September 1, 2025, and September 1, 2026. Before the stress ball application after open heart surgery, participants in the control and study groups will be asked to complete the Descriptive Characteristics Form, VAS, VAS-A, and Hemodynamic Variables Monitoring Form. The Hemodynamic Variables Monitoring Form will be completed by the researcher (F.E.Ö) while monitoring the patient on the bedside monitor (Nihon Kohden, Tokyo). Participants who complete the Descriptive Characteristics Form,
  The control group will not receive any treatment other than routine treatment and will be evaluated at the same time as the study group.
- Stress ball group (Experimental): In addition to the clinic's routine treatment and care, patients in the study group will be treated with a stress ball during chest tube removal. 15 minutes before the procedure, nurses (FEÖ and NT) will explain and demonstrate how to use the stress ball. The stress ball application will last approximately five minutes, including the chest tube removal procedure. A round, medium-hard, high-quality silicone ball, approximately 6 cm in diameter, will be used. Patients will be asked to hold the ball in their palms, count to three, squeeze, and release once. Patients will be instructed to continue this exercise until the chest tube removal procedure is complete, and then, under the supervision of the researcher, for an average of five minutes, focusing their attention on the stress ball. The ball will be washed and cleaned after each use and wiped with disposable asepsis wipes before being administered to the patient. The control group will not receive any other treatment beyond routine t
  Interventions: Other: Stress ball

INTERVENTIONS:
Other: Stress ball — Recently, the use of non-pharmacological methods applied by nurses has become increasingly widespread. One independent nursing practice for reducing pain and anxiety is the stress ball. A stress ball, one of these non-pharmacological methods, utilizes the sense of touch to divert attention and cognitive focus. This simple, reliable, and low-cost method reduces pain and anxiety by directing the mind to a salient stimulus.
  Arms: Stress ball group

SUMMARY:
15 minutes before the procedure, nurses (FEÖ and NT) will explain and demonstrate how to use the stress ball. The stress ball will be applied for approximately five minutes, including the chest tube removal procedure. A round, medium-hard, high-quality silicone ball, approximately 6 cm in diameter, will be used. Patients will be asked to hold the ball in their palms, count to three, squeeze, and release once. Patients will be instructed to continue this exercise until the chest tube removal procedure is completed, and then, under the supervision of the researcher, for approximately five minutes, focusing their attention on the stress ball. The ball will be washed and cleaned after each use and wiped with disposable asepsis wipes before being administered to the patient. The control group will not receive any other treatment beyond routine treatment and will be assessed at the same time as the study group.

The chest tube will be removed by a physician during the stress ball application. Procedural pain level, anxiety level and hemodynamic variables of all patients in the study and control groups will be re-evaluated immediately after chest tube removal and 15 and 30 minutes after chest tube removal.

DETAILED DESCRIPTION:
Chest tubes are routinely removed on the second or third postoperative day in patients in the Cardiovascular Surgery Intensive Care Unit, and patients with stable hemodynamic variables are discharged to the clinic. Morphine (0.01 mg) and paracetamol (if necessary) are used for routine analgesic treatment during the intensive care unit. Data will be collected between September 1, 2025, and September 1, 2026. Before the stress ball application after open heart surgery, participants in the control and study groups will be asked to complete the Descriptive Characteristics Form, VAS, VAS-A, and Hemodynamic Variables Monitoring Form. The Hemodynamic Variables Monitoring Form will be completed by the researcher (F.E.Ö) while monitoring the patient on the bedside monitor (Nihon Kohden, Tokyo). Participants who complete the Descriptive Characteristics Form, VAS, and VAS-A, and whose hemodynamic parameters are recorded, will be administered the stress ball application by Firdevs Ebru Özdemir and Nesrin Temiz.In addition to the clinic's routine treatment and care, patients in the study group will receive a stress ball during chest tube removal. 15 minutes before the procedure, nurses (FEÖ and NT) will explain and demonstrate how to use the stress ball. The stress ball will be applied for approximately five minutes, including the chest tube removal procedure. A round, medium-hard, high-quality silicone ball, approximately 6 cm in diameter, will be used. Patients will be asked to hold the ball in their palms, count to three, squeeze, and release once. Patients will be instructed to continue this exercise until the chest tube removal procedure is completed, and then, under the supervision of the researcher, for approximately five minutes, focusing their attention on the stress ball. The ball will be washed and cleaned after each use and wiped with disposable asepsis wipes before being administered to the patient. The control group will not receive any other treatment beyond routine treatment and will be assessed at the same time as the study group.

The chest tube will be removed by a physician during the stress ball application. Procedural pain level, anxiety level and hemodynamic variables of all patients in the study and control groups will be re-evaluated immediately after chest tube removal and 15 and 30 minutes after chest tube removal.

ELIGIBILITY:
Inclusion Criteria:Patients will be included : have only one chest tube after open heart surgery,

* are 18 years of age or older,
* are conscious and cooperative,
* speak and understand Turkish,
* have a stable general condition and hemodynamic variables,
* have a planned surgical procedure,
* have no previous chest tube experience,
* have no psychiatric diagnosis,
* are not using psychiatric and/or local neuromuscular blocking medications,
* agree to participate in the study (sign the Informed Consent Form).

Exclusion Criteria:Patients who do not have a chest tube or have multiple chest tubes after open heart surgery,

* Are under 18 years of age,
* Are conscious and uncooperative,
* Do not speak or understand Turkish,
* Are in an unstable general condition or hemodynamic variables,
* Have undergone emergency surgery,
* Have previous chest tube placement experience,
* Have a current psychiatric diagnosis,
* Are taking psychiatric and/or local neuromuscular blocking medications,
* Do not agree to participate in the study (do not sign the Informed Consent Form) will not be included in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2025-11-27 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-06-20 (Estimated)

PRIMARY OUTCOMES:
Participants' pain levels with stress ball application | Before, immediately after, 15 minutes and 30 minutes after chest tube removal
  Visual Analog Scale (VAS): Developed by Freyd (1923), the VAS is a single, 10-cm-long scale that can be used vertically or horizontally to assess pain levels. A generally accepted, reliable, and easily applicable scale, the VAS consists of a 10-cm-long line with subjective descriptive statements at either end of the scale (0 cm = none at all and 10 cm = maximum presence). The individual places a mark on this 10-cm line at the appropriate location on the scale. The distance from the beginning of the scale to the mark is measured with a ruler, and the individual's pain level is numerically determined in cm.

SECONDARY OUTCOMES:
anxiety | Before, immediately after, 15 minutes and 30 minutes after chest tube removal
  The VAS-A was developed to convert numerical values that cannot be measured numerically. A generally accepted, reliable, and easily applicable measurement tool in the world literature, the VAS consists of a 10-cm-long line with subjective descriptive statements at either end (0 cm = not present at all and 10 cm = most present). Research has shown that the VAS-A has been used to assess anxiety in patients before surgical interventions. Individuals place a mark at the appropriate location on this 10-cm line. The distance from the beginning of the scale to the mark is measured with a ruler, and the individual's anxiety level is numerically determined in cm. A low score on the VAS-A indicates a low/mild anxiety level, while a high score indicates a high/severe anxiety level.
Systolic blood pressure changes after stress ball | Before, immediately after, 15 minutes and 30 minutes after chest tube removal
  This form will record the systolic blood pressure, diastolic blood pressure, heart rate, respiratory rate, and oxygen saturation values of the study and control groups measured at the specified times. Hemodynamic variables will be monitored and recorded using a bedside monitor (Nihon Kohden, Tokyo). To ensure data reliability and accuracy, these monitors are calibrated monthly by the biomedical engineering department, in accordance with hospital policy.
Diastolic blood pressure changes after stress ball | Before, immediately after, 15 minutes and 30 minutes after chest tube removal
  This form will record the systolic blood pressure, diastolic blood pressure, heart rate, respiratory rate, and oxygen saturation values of the study and control groups measured at the specified times. Hemodynamic variables will be monitored and recorded using a bedside monitor (Nihon Kohden, Tokyo). To ensure data reliability and accuracy, these monitors are calibrated monthly by the biomedical engineering department, in accordance with hospital policy.
Heart rate changes after stress ball | Before, immediately after, 15 minutes and 30 minutes after chest tube removal
  This form will record the systolic blood pressure, diastolic blood pressure, heart rate, respiratory rate, and oxygen saturation values of the study and control groups measured at the specified times. Hemodynamic variables will be monitored and recorded using a bedside monitor (Nihon Kohden, Tokyo). To ensure data reliability and accuracy, these monitors are calibrated monthly by the biomedical engineering department, in accordance with hospital policy.
Respiratory rate changes after stress ball | Before, immediately after, 15 minutes and 30 minutes after chest tube removal
  This form will record the systolic blood pressure, diastolic blood pressure, heart rate, respiratory rate, and oxygen saturation values of the study and control groups measured at the specified times. Hemodynamic variables will be monitored and recorded using a bedside monitor (Nihon Kohden, Tokyo). To ensure data reliability and accuracy, these monitors are calibrated monthly by the biomedical engineering department, in accordance with hospital policy.
Oxygen saturation values changes after stress ball | Before, immediately after, 15 minutes and 30 minutes after chest tube removal
  This form will record the systolic blood pressure, diastolic blood pressure, heart rate, respiratory rate, and oxygen saturation values of the study and control groups measured at the specified times. Hemodynamic variables will be monitored and recorded using a bedside monitor (Nihon Kohden, Tokyo). To ensure data reliability and accuracy, these monitors are calibrated monthly by the biomedical engineering department, in accordance with hospital policy.

CONTACTS AND LOCATIONS:
Locations (1):
- Turkey, Mersin University,, Yenişehir, Mersin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Yarahmadi S, Mohammadi N, Ardalan A, Najafizadeh H, Gholami M. The combined effects of cold therapy and music therapy on pain following chest tube removal among patients with cardiac bypass surgery. Complement Ther Clin Pract. 2018 May;31:71-75. doi: 10.1016/j.ctcp.2018.01.006. Epub 2018 Feb 6. PMID 29705484